CLINICAL TRIAL: NCT03558399
Title: A Randomized Controlled Trial Comparing Live Birth From Single, Euploid Frozen Blastocyst Transfer Using Conventional Timing Versus Timing by Endometrial Receptivity Analysis
Brief Title: Frozen Blastocyst Transfer Using Conventional Timing Versus Timing by Endometrial Receptivity Analysis
Acronym: Synchrony
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shady Grove Fertility Reproductive Science Center (Other)
Collaborators: Igenomix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 1183343
Record Dates: First submitted 2018-04-25; First posted 2018-06-15 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Implantation Failure; Infertility, Female
Keywords: Endometrial receptivity analysis; Window of implantation; Euploid; Infertility, Female; Implantation failure; Frozen embryo transfer FET; ERA; WOI; FET; Synchrony
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Results of the ERA analysis will not be disclosed to the patient or the physician or the outcome assessor, nor will the study arm to which the patient was assigned, though the patient/physician may be able to intuit assignment to the ERA arm based on the frozen embryo transfer time that she is assigned. The date and time of embryo transfer will be provided by the investigator/research team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FET according to ERA (Experimental): In preparation for frozen embryo transfer (FET), estradiol will be administered for approximately 10 to 14 days or until endometrial criteria are met. These endometrial criteria will be assessed with transvaginal ultrasound and serum estradiol levels. Women will then begin intramuscular progesterone injection and if assigned to the study arm, a single euploid embryo will be transferred at the time indicated by the ERA test results. Merely the timing of embryo transfer will distinguish the study from the control group.
  Interventions: Other: FET according to ERA
- FET according to standard protocol (Active Comparator): In preparation for frozen embryo transfer (FET), estradiol will be administered for approximately 10 to 14 days or until endometrial criteria are met. These endometrial criteria will be assessed with transvaginal ultrasound and serum estradiol levels. Women will then begin intramuscular progesterone injection and if assigned to the control arm, a single euploid embryo will be transferred according to our standard FET protocol.
  Interventions: Other: FET according to standard protocol

INTERVENTIONS:
Other: FET according to ERA — Single euploid FET will be performed at the time indicated by the ERA test results.
  Arms: FET according to ERA
Other: FET according to standard protocol — Single euploid FET will be performed according to our standard FET protocol.
  Arms: FET according to standard protocol

SUMMARY:
To assess live birth after embryo transfer according to an individual's ERA results as opposed to routine protocol for frozen embryo transfer (FET) cycles.

DETAILED DESCRIPTION:
It has been proposed, that the receptivity status of the endometrium shifts among individual women and that repeated implantation failure is ascribable to an endometrial factor in up to 25%. The endometrial receptivity analysis (ERA) is a diagnostic method that was developed based on the unique genomic signature of the endometrium during the window of implantation and classifies the endometrium as receptive, pre-receptive or post-receptive to guide embryo transfer.

The purpose of this assessor-blind, randomized clinical study is to determine whether live birth from vitrified/thawed euploid embryo transfer is improved when transfer is timed according to endometrial receptivity analysis (ERA) results.

Approximately 800 women (n=400 in each arm) will be enrolled according to the inclusion/exclusion criteria among patients of Shady Grove Fertility. Participants will undergo a standard in vitro fertilization (IVF) cycle, followed by preimplantation genetic screening (PGS) provided a high quality blastocyst is available. Participants with at least one PGS normal (euploid) embryo will be randomized (assigned by chance, like the flip of a coin) to one of two study groups. Women in both study arms will then undergo ERA testing and neither the patients nor their treating physicians will know to which group the women have been assigned to, or the ERA testing results. Up until this point there is no difference between the study and control group. The investigational aspect of this trial is described as follows: If the participant is assigned to the study arm, the single, euploid, frozen embryo transfer (FET) during the subsequent cycle will be performed at the time indicated by the ERA test results. If she is in the control arm, the embryo will be transferred according to our standard FET protocol.

Patients enrolling in the study will receive PGS and ERA free of charge.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Female age between 30 and 40 years and deemed likely by her physician, based on ovarian reserve testing, to produce at least one euploid blastocyst via one IVF/intracytoplasmatic sperm injection (ICSI) cycle
3. Having ≥ 1 euploid embryo available for embryo transfer
4. Standard eligibility criteria to undergo IVF and FET at Shady Grove Fertility Center.

Exclusion Criteria:

1. Known uterine factor impacting the endometrium
2. Use of surgically aspirated sperm for fertilization
3. Presence of any clinically relevant systemic disease that contraindicates assisted reproductive technology.
4. Since the subject last had a live birth (if any), there have been more than two embryo transfers that have not resulted in ongoing pregnancy
5. Body mass index >40 kg/m2 at screening
6. Recurrent pregnancy loss, defined as two or more clinical pregnancy losses without live birth
7. Planned testing of embryos for single gene disorder(s) or structural chromosome rearrangements
8. Currently breast feeding, pregnant, or contraindication to pregnancy

Ages: 30 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only biological female subjects will be recruited for this study as an evaluation of the endometrium requires a uterus to be present and therefore this is only possible in the biological female sex.
Enrollment: 800 (Estimated)
Dates: Start 2018-04-25 (Actual); Primary Completion 2021-09-23 (Estimated); Study Completion 2021-09-23 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure of this clinical trial is to assess live birth after euploid embryo transfer according to an individual's ERA result as opposed to routine protocol for frozen embryo transfer (FET) cycles. | From date of randomization until live born infant at an estimated gestational age of at least 23 weeks or greater

SECONDARY OUTCOMES:
A secondary outcome measure of this clinical trial is to assess ongoing implantation rate after embryo transfer according to an individual's ERA result as opposed to routine protocol for frozen embryo transfer (FET) cycles. | From date of randomization until 7-8 weeks estimated gestational age
  The ongoing implantation rate is defined as maximum number of fetal heartbeats divided by total number of embryos transferred
A secondary outcome measure of this clinical trial is to assess implantation rate after embryo transfer according to an individual's ERA result as opposed to routine protocol for frozen embryo transfer (FET) cycles. | From date of randomization until 5-6 weeks estimated gestational age
  The implantation rate is defined as the maximum number of gestational sacs per patient
A secondary outcome measure of this clinical trial is to assess biochemical pregnancy after embryo transfer according to an individual's ERA result as opposed to routine protocol for frozen embryo transfer (FET) cycles. | From date of randomization until ~10 days following embryo transfer
  Biochemical pregnancy is defined as detection of beta hCG above 5 IU/L
A secondary outcome measure of this clinical trial is to assess clinical pregnancy after embryo transfer according to an individual's ERA result as opposed to routine protocol for frozen embryo transfer (FET) cycles. | From date of randomization until 5-7 weeks estimated gestational age
  The clinical pregnancy rate is defined as the presence of gestational sacs

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Devine, MD, Principal Investigator — Shady Grove Fertility
Locations (1):
- Shady Grove Fertility Reproductive Science Center, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruiz-Alonso M, Blesa D, Diaz-Gimeno P, Gomez E, Fernandez-Sanchez M, Carranza F, Carrera J, Vilella F, Pellicer A, Simon C. The endometrial receptivity array for diagnosis and personalized embryo transfer as a treatment for patients with repeated implantation failure. Fertil Steril. 2013 Sep;100(3):818-24. doi: 10.1016/j.fertnstert.2013.05.004. Epub 2013 Jun 4. PMID 23756099
- [Background] Katzorke N, Vilella F, Ruiz M, Krussel JS, Simon C. Diagnosis of Endometrial-Factor Infertility: Current Approaches and New Avenues for Research. Geburtshilfe Frauenheilkd. 2016 Jun;76(6):699-703. doi: 10.1055/s-0042-103752. PMID 27365540
- [Background] Horcajadas JA, Pellicer A, Simon C. Wide genomic analysis of human endometrial receptivity: new times, new opportunities. Hum Reprod Update. 2007 Jan-Feb;13(1):77-86. doi: 10.1093/humupd/dml046. Epub 2006 Sep 7. PMID 16960016
- [Background] Ponnampalam AP, Weston GC, Trajstman AC, Susil B, Rogers PA. Molecular classification of human endometrial cycle stages by transcriptional profiling. Mol Hum Reprod. 2004 Dec;10(12):879-93. doi: 10.1093/molehr/gah121. Epub 2004 Oct 22. PMID 15501903
- [Background] Galliano D, Pellicer A. MicroRNA and implantation. Fertil Steril. 2014 Jun;101(6):1531-44. doi: 10.1016/j.fertnstert.2014.04.023. PMID 24882617
- [Background] Ruiz-Alonso M, Blesa D, Simon C. The genomics of the human endometrium. Biochim Biophys Acta. 2012 Dec;1822(12):1931-42. doi: 10.1016/j.bbadis.2012.05.004. Epub 2012 May 24. PMID 22634130
- [Derived] Doyle N, Jahandideh S, Hill MJ, Widra EA, Levy M, Devine K. Effect of Timing by Endometrial Receptivity Testing vs Standard Timing of Frozen Embryo Transfer on Live Birth in Patients Undergoing In Vitro Fertilization: A Randomized Clinical Trial. JAMA. 2022 Dec 6;328(21):2117-2125. doi: 10.1001/jama.2022.20438. PMID 36472596